CLINICAL TRIAL: NCT03035461
Title: Ressenti du Patient au Moment de l'Annonce du Diagnostic de DMLA
Brief Title: Patient's Feelings After Receiving a Diagnosis of Age-related Macular Degeneration
Acronym: PANDA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Principal Investigator, Joëlle Marciano, Orthoptist in the ophtalmologic department of the CHI Creteil, Centre Hospitalier Intercommunal Creteil
Other Study IDs: PANDA
Record Dates: First submitted 2017-01-25; First posted 2017-01-30 (Estimated); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Age Related Macular Degeneration
Keywords: diagnosis annoucement; patient's feelings
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Age-related macular degeneration (AMD) is the leading cause of blindness in the elderly population of the industrialized world. AMD is a progressive degenerative disease affecting the central area of the retina, responsible for distinct vision. Vision loss arises from aberrant new vessel growth which causes the accumulation of blood or fluid within the retina's thickness and eventually leads to permanent scarring. The two major forms of AMD are exudative, or neovascular or "wet", and non-exudative, or "dry".

Vascular endothelial growth factor (VEGF) represents the key modulator of the angiogenetic process and is involved in the pathophysiology of AMD. Anti VEGF therapies are used to treat wet-AMD.

After diagnosis and explanations of the practionner, the patients and their close relatives have still frequently many questions about the intravitreal injections, the prognosis, the risk of visual impairment, etc. Few teams have studied the modalities of diagnosis announcement and the understanding of the patients on the disease course.

The aim of this study is to evaluate the feelings after the AMD diagnosis announcement as well as the understanding of the possibilities of treatment and the clinical surveillance.

ELIGIBILITY:
Inclusion Criteria:

* patient up to 55 years old
* wet AMD
* diagnostic questionnaire group: patient being announced with AMD for less than 1 month
* disease course questionnaire group: patients treated by anti-VEGF from 6 to 12 months

Exclusion Criteria:

* dry AMD
* patient under 55 years old
* patient who doesn't speak French
* patient carrying an ophtalmologic genetic disorder

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of wet AMD seen in the ophtalmologic department of the CHI creteil
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
Description of the patient's feelings | up to 1 month after diagnosis
  A questionnaire with a list of different feelings: anxiety, distress, relief, resigned, guilty, etc. is proposed to the patient after AMD diagnosis. they can also explain their feelings by themselves.

SECONDARY OUTCOMES:
score of general satisfaction | up to 1 month after diagnosis
  the patient will score their satisfaction on a numeric scale from 0 (not satisfied at all) to 10 (extremely satisfied)
score on a comprehension quiz on AMD | up to 1 month after diagnosis
Score on a composite score evaluating the clarity of medical explanations | up to 1 month after diagnosis
Score on a composite score evaluating the clarity of medical explanations | between 6 months and 1 year of follow-up
score of satisfaction of announcement conditions | up to 1 month after diagnosis
score of satisfaction of announcement conditions | between 6 months and 1 year of follow-up
score of satisfactions regarding the clarity of the disease course and treatment explanations | between 6 months and 1 year of follow-up
Score on the anxiety PHQ9 questionnaire | between 6 months and 1 year of follow-up
Score on the anxiety GAD7 questionnaire | between 6 months and 1 year of follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Marciano Joelle, Créteil, Creteil, France

IPD SHARING:
Plan to Share IPD: No